CLINICAL TRIAL: NCT02248818
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses of AZD8108 in Healthy Volunteers
Brief Title: AZD8108 SAD/MAD in Healthy Volunteers
Acronym: AZD8108
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D5800C00001
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZD8108 (Experimental): Subjects will participate in 1 of 7 groups and receive single or multiple doses of AZD8108 or matching placebo. In each group 6 subjects will receive AZD8108
  Interventions: Drug: AZD8108
- Placebo to match AZD8108 (Placebo Comparator): Subjects will participate in 1 of 7 groups and receive single or multiple doses of AZD8108 or matching placebo. In each group 2 subjects will receive matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8108 — Drug: AZD8108 Single or Multiple doses administered orally as a solution.
  Arms: AZD8108
Drug: Placebo — Placebo to match AZD8108 Single or Multiple doses of matching placebo administered orally as a solution
  Arms: Placebo to match AZD8108

SUMMARY:
This is a randomized, double-blind, placebo-controlled study of single and multiple ascending dosage levels of AZD8108 in healthy volunteers. The study includes an up to 28-day screening period, an in-house period during which AZD8108 or placebo will be administered orally as a solution, and a 4- to 10-day follow-up period after discharge.

DETAILED DESCRIPTION:
In Part 1 of the study (single ascending dose portion), approximately 32 subjects will be randomly assigned. Eight (8) subjects will be randomized in each of 4 dosage-level cohorts (AZD8108 or placebo). Within each cohort, 6 subjects will be randomized to receive AZD8108 and 2 subjects will be randomized to receive placebo. Each subject will receive only one dose of either AZD8108 or placebo on Day 1. In Part 2 of the study (multiple ascending dose portion), approximately 24 subjects will be randomly assigned. Eight (8) subjects will be randomized in each of 3 dosage-level cohorts. Within each cohort, 6 subjects will be randomized to receive AZD8108 and 2 subjects will be randomized to receive placebo. Each subject will receive twelve doses of either AZD8108 or placebo

ELIGIBILITY:
Inclusion Criteria: Inclusion Criteria: 1. Subjects must understand the nature of the study and must provide signed and dated written informed consent in accordance with local regulations before the conduct of any study-specific procedures. 2. Men and postmenopausal or surgically sterile women age 18-55 years inclusive. 3. Subjects must have a body mass index (BMI) between 19 and 30, inclusive and weigh between 50kg and 100kg inclusive. 4.Subjects must be fluent in English.

-

Exclusion Criteria:1. A history or presence of a clinically significant hepatic, renal, gastrointestinal, cardiovascular, endocrine, respiratory, immunologic, hematologic, dermatologic, or neurologic abnormality. 2. A clinically significant abnormality on physical examination, neurological examination, EEG, ECG, vital signs or laboratory evaluations at screen or between screen and dose administration. 3. A history of seizure. 4.A history of head trauma, including closed head injury with loss of consciousness. 5.Any history of suicide attempt or suicidal behavior, or, in the opinion of the investigator, clinically significant risk of suicide or violent behavior. 6. Urine drug screen positive for a drug of abuse 7. A family history of schizophrenia, schizoaffective disorder, or psychosis in first degree relatives.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 258 (Actual)
Dates: Start 2014-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mina Pastagia, MD, MS, Principal Investigator — Clinilabs, Inc.
Locations (1):
- Clinilabs, Inc., New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy Adult volunteer study, Part 1: SAD: single ascending dose cohorts, followed by Part 2: MAD: multiple ascending dose cohorts. Plan was for each cohort to have 8 subjects, 2 placebo dosed and 6 AZD8108 dosed.
Pre-assignment Details: Protocol allowed for 258 subjects to be screened, only 155 subjects were screened before all cohorts for the study were filled and recruitment ended.
Groups:
- AZD8108 20 mg SAD: AZD8108 20 mg SAD, Cohort 1
- AZD8108 60 mg SAD: AZD8106 60 mg SAD, Cohort 2
- AZD8108 95 mg SAD: AZD8108 95 mg SAD, Cohort 3
- Placebo SAD: Placebo SAD, pooled across Cohorts 1 - 3
- AZD8108 50 mg: AZD8108 50 mg MAD, Cohort 5
- AZD8108 90 mg MAD (6): AZD8108 90 mg MAD, Cohort 6
- AZD8108 90 mg MAD (7): AZD8108 90 mg MAD, Cohort 7
- Placebo MAD: Placebo MAD, pooled across Cohorts 5 & 7
- Screen: Screen - no treatment
Period: Screening
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD | Screen
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 155
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 48
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 107
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Not completed — Study fully enrolled | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 73
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Period: Randomised Study
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD | Screen
Started | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 4 | 0
Completed | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 4 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0
Not completed — Administrative - randomization error | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AZD8108 20 mg - SAD: AZD8108 20 mg SAD, Cohort 1
- AZD8108 60 mg - SAD: AZD8108 60 mg SAD, Cohort 2
- AZD8108 95 mg - SAD: AZD8108 95 mg SAD, Cohort 3
- AZD8108 50 mg MAD: AZD8108 50 mg MAD, Cohort 5
- Total: Total of all reporting groups
Arm/Group | AZD8108 20 mg - SAD | AZD8108 60 mg - SAD | AZD8108 95 mg - SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 4 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.0 (10.81) | 36.3 (12.55) | 38.7 (10.53) | 38.0 (10.53) | 36.7 (7.89) | 35.4 (10.31) | 31.2 (2.64) | 39.3 (9.22) | 36.0 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  Male | 4 | 6 | 6 | 5 | 6 | 8 | 6 | 4 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 2 | 2 | 5 | 0 | 1 | 13
  Not Hispanic or Latino | 4 | 6 | 5 | 4 | 4 | 3 | 5 | 2 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 3 | 3 | 2 | 2 | 3 | 2 | 21
  White | 2 | 2 | 2 | 1 | 1 | 3 | 3 | 1 | 15
  More than one race | 2 | 0 | 1 | 2 | 2 | 2 | 0 | 1 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety Laboratory - Thyroid Stimulating Hormone Above Upper Limit of Normal
Description: Safety Laboratory - Thyroid Stimulating Hormone participants with laboratory value above the upper limit of normal
Time Frame: Day -1 to 7 days after last dose
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 4
Participants | 2 | 3 | 0 | 0 | 4 | 3 | 0 | 0

2. Primary Outcome: Pharmacokinetic :Area Under the Concentration Curve (0 to Infinity), AZD6765 After Single/1st Dose of AZD8108
Description: Pharmacokinetic : Area under the concentration curve (0 to infinity), AZD6765 after single/first dose of AZD8108
Time Frame: Pre-dose,5,15,30 min, 1,1.5,2,3,4,6,8,10,12,14,16,24,48,(72 SAD only) hr after day 1 dose
Population: Pharmacokinetic Population (those dosed with AZD8108)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 8 | 6 | 0
hours*ng/mL | 726 (22.4) | 2651 (17.1) | 4533 (11.3) |  | 2160 (37.8) | 4318 (13.2) | 4597 (21.8) |

3. Primary Outcome: Pharmacokinetic :Area Under the Concentration Curve (0 to 24 Hour), AZD6765 MAD Day 6 Dose of AZD8108
Description: Pharmacokinetic : Area under the concentration curve (0 to 24 hour), AZD6765 MAD Day 6 dose of AZD8108 Cohort 5 & 7, Cohort 6 did not reach Day 6
Time Frame: Pre-dose, 5,15,30 min, 1,1.5,2,3,4,6,8,10,12,16,24 hr after Day 6 dose
Population: Pharmacokinetic Population (those dosed with AZD8108)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 6 | 0
hours*ng/mL |  |  |  |  | 2061 (34.7) |  | 4408 (26.3) |

4. Primary Outcome: Pharmacokinetic :Area Under the Concentration Curve (0 to Infinity), AZD6765 MAD Day 12 Dose of AZD8108
Description: Pharmacokinetic : Area under the concentration curve (0 to infinity), AZD6765 MAD Day 12 dose of AZD8108 Cohort 5 & 7, Cohort 6 did not reach Day 12
Time Frame: Pre-dose, 5,15,30 min, 1,1.5,2,3,4,6,8,10,12,16,24,48, 72 hr after Day 12 dose
Population: Pharmacokinetic Population (those dosed with AZD8108)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 6 | 0
hours*ng/mL |  |  |  |  | 2837 (47.6) |  | 6733 (30.2) |

5. Primary Outcome: Pharmacokinetic :Area Under the Concentration Curve (0 to 24 Hours), AZD6765 After DAY 12 Dose of AZD8108
Description: Pharmacokinetic : Area under the concentration curve (0 to 24 hours), AZD6765 after Day 12 dose of AZD8108 cohort 5 & 7, Cohort 6 dod not reach Day 12
Time Frame: Pre-dose, 5,15,30 min, 1,1.5,2,3,4,6,8,10,12,16, and 24 hours after dose
Population: Pharmacokinetic Population (those dosed with AZD8108)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 6 | 0
hours*ng/mL |  |  |  |  | 2191 (38.1) |  | 4670 (20.7) |

6. Primary Outcome: Pharmacokinetic : Maximum Concentration of AZD6765 After Single/1st Dose of AZD8108
Description: Pharmacokinetic : Maximum concentration of AZD6765 after single/first dose of AZD8108
Time Frame: Pre-dose, 5,15,30 min, 1,1.5,2,3,4,6,8,10,12,16,25,48,972 SAD only)hr after Day 1 dose
Population: Pharmacokinetic Population (those dosed with AZD8108)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 8 | 6 | 0
ng/mL | 50.1 (22.4) | 148 (19.3) | 264 (17.8) |  | 146 (27.5) | 287 (22.7) | 236 (10.6) |

7. Primary Outcome: Pharmacokinetic : Maximum Concentration of AZD6765 After MAD Day 6 Dose of AZD8108
Description: Pharmacokinetic : Maximum concentration of AZD6765 after MAD Day 6 dose of AZD8108, Cohorts 5 & 7, Cohort 6 did not reach Day 6
Time Frame: Pre-dose, 5,15.30 min, 1,1.5,2,3,4,6,8,10,12,16,24 hr after Day 6 dose
Population: Pharmacokinetic Population (those dosed with AZD8108) MAD cohorts 5 & 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 6 | 0
ng/mL |  |  |  |  | 176 (23.9) |  | 330 (18.7) |

8. Primary Outcome: Pharmacokinetic : Maximum Concentration of AZD6765 After MAD Day 12 Dose of AZD8108
Description: Pharmacokinetic : Maximum concentration of AZD6765 after MAD Day 12 dose of AZD8108, Cohorts 5 & 7, Cohort 6 did not reach Day 12
Time Frame: Pre-dose, 5,15,30 min, 1,1.5,2,3,4,6,8,10,12,16,24,48,72 hr after Day 12 dose
Population: Pharmacokinetic Population (those dosed with AZD8108) MAD cohorts 5 & 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 6 | 0
ng/mL |  |  |  |  | 197 (30.4) |  | 337 (11.3) |

9. Secondary Outcome: Pharmacokinetic: Time to Maximum Plasma Concentration of AZD6765 After Single (SAD)/ 1st (MAD) Dose of AZD8108
Description: Pharmacokinetic: Time to Maximum plasma concentration of AZD6765 after single (SAD) / first (MAD) dose AZD8108
Time Frame: Pre-dose, 5,15,30 min, 1,1.5,2,3,4,6,8,10,12,16,24,48,(72 SAD only) hr after day 1 dose
Population: Pharmacokinetic population (subjects dosed with AZD8108)
Measure: Median (Full Range); unit: hours
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 8 | 6 | 0
hours | 1.75 [1.00 to 3.03] | 2.00 [1.00 to 3.00] | 2.50 [1.00 to 6.00] |  | 1.25 [1.00 to 4.00] | 1.28 [1.00 to 3.00] | 2.55 [1.52 to 10.00] |

10. Secondary Outcome: Pharmacokinetic: Fraction of Equivalent Dose of AZD6765 Excreted in Urine (SAD) After Single Dose of AZD8108
Description: Pharmacokinetic: Fraction of equivalent dose of AZD6765 excreted in urine (SAD) after single dose of AZD8108 (Cohorts 1 - 3)
Time Frame: Collection 0-6, 6-12,12-24, 24-48, (48-72 SAD only) hy after Day 1 dose
Population: Pharmacokinetic Population (Cohorts 1-3) AZD8108 dosed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent
Units Other Than Participants: Participants with urine volume data
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0
Number analyzed (Participants with urine volume data) | 5 | 6 | 5 | 0 | 0 | 0 | 0 | 0
Percent | 48.8 (55.2) | 33.8 (30.1) | 38.8 (8.24) |  |  |  |  |

11. Secondary Outcome: Pharmacokinetic: Fraction of Equivalent Dose of AZD6765 Excreted in Urine (MAD) After Day 12 Dose of AZD8108
Description: Pharmacokinetic: Fraction of equivalent dose of AZD6765 excreted in urine (MAD) after Day 12 dose of AZD8108 Cohorts 5 & 7, Cohort 6 did not reach day 12
Time Frame: Collection 0-6, 0-12, 12-24, 24-48, 48-72 hr after Day 12 dose
Population: Pharmacokinetic Population (Cohorts 1-3) AZD8108 dosed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 6 | 0
Percent |  |  |  |  | 49.4 (28.1) |  | 30.2 (35.5) |

12. Secondary Outcome: Pharmacokinetic: Time to Maximum Plasma Concentration of AZD6765 After Day 12 (MAD) Dose of AZD8108
Description: Pharmacokinetic: Time to Maximum plasma concentration of AZD6765 after Day 12 (MAD) dose AZD8108 Cohorts 5 & 7, Cohort 6 did not reach day 12
Time Frame: Pre-dose, 5,15,30 min, 1,1.5,2,3,4,6,8,10,12,16,24,48,72 hours after Day 12 dose
Population: Pharmacokinetic population (subjects dosed with AZD8108)
Measure: Median (Full Range); unit: hours
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 6 | 0
hours |  |  |  |  | 1.75 [0.50 to 2.00] |  | 1.80 [1.00 to 3.00] |

13. Secondary Outcome: Pharmacokinetic: Accumulation Index for Area Under Concentration Curve (0 to 24 Hour) MAD
Description: Pharmacokinetic: Accumulation index for Area Under Concentration Curve (0 to 24 hour) MAD Cohorts 5 & 7, cohort 6 did not reach day 12 [accumulation index (Day 6 or 12 /Day1)]
Time Frame: Day 12 compared to Day 1
Population: Pharmacokinetic population, MAD Cohorts 5 & 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 6 | 0
ratio
  Day 6 |  |  |  |  | 1.30 (0.181) |  | 1.37 (0.224) |
  Day 12 |  |  |  |  | 1.39 (0.254) |  | 1.44 (0.165) |

14. Other Pre Specified Outcome: EEG Parameter (DAY 1) - Gamma - Change From Baseline in Total Area of the Brain (Eyes Closed)- Consistent Change in Either Direction
Description: EEG parameter (DAY 1) - Gamma - Change from baseline in Total Area of the Brain (eyes closed) - to identify a dose related change in EEG gamma bands to assess target engagement, a consistent change in either direction relative to placebo would be of interest
Time Frame: 8 hours after dose
Population: Safety population
Measure: Mean (Standard Deviation); unit: uV2
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 4
uV2
  0.5 hours after dose | -0.069 (0.3715) | -0.272 (0.2422) | -0.166 (0.1880) | .0141 (0.2358) | -0.343 (0.3348) | 0.087 (0.3979) | -0.154 (0.2555) | 0.128 (0.5069)
  1 hour after dose | 0.101 (0.2638) | -0.238 (0.4504) | -0.140 (0.2520) | -0.003 (0.1467) | -0.109 (0.5843) | 0.092 (0.3466) | -0.063 (0.2291) | -0.121 (0.2005)
  1.5 hours after dose | -0.113 (0.2616) | -0.161 (0.6017) | -0.069 (0.2095) | 0.097 (0.3402) | 0.211 (0.5514) | -0.052 (0.3888) | 0.016 (0.3687) | 0.313 (0.2701)
  2 hours after dose | 0.244 (0.2577) | -0.347 (0.3231) | -0.080 (0.2324) | -0.086 (0.2350) | -0.303 (0.4675) | -0.142 (0.2639) | -0.097 (0.2185) | 0.019 (0.2661)
  3 hours after dose | 0.214 (0.2120) | -0.254 (0.2461) | -0.108 (0.1569) | 0.126 (0.1181) | -0.369 (0.4360) | 0.058 (0.4186) | 0.011 (0.3292) | 0.247 (0.4936)
  5 hours after dose | -0.225 (0.1615) | -0.454 (0.2641) | -0.014 (0.1025) | 0.138 (0.3071) | -0.514 (0.4117) | -0.073 (0.3506) | -0.25 (0.2971) | -0.151 (0.2954)
  8 hours after dose | 0.222 (0.5150) | -0.263 (0.1219) | -0.086 (0.3075) | 0.091 (0.4193) | -0.125 (0.4958) | -0.169 (0.3217) | -0.124 (0.3209) | 0.034 (0.3623)

15. Other Pre Specified Outcome: EEG Parameter (DAY 6) - Gamma - Change From Baseline in Total Area of the Brain (Eyes Closed)- Consistent Change in Either Direction
Description: EEG parameter (DAY 6) - Gamma - Change from baseline in Total Area of the Brain (eyes closed) Cohort 5 & 7, Cohort 6 did not reach Day 6; to identify a dose related change in EEG gamma bands to assess target engagement, a consistent change in either direction compared to placebo was of interest
Time Frame: 8 hours after dose
Population: Safety population
Measure: Mean (Standard Deviation); unit: uV2
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 6 | 4
uV2
  Pre-dose Day 6 dose |  |  |  |  | -0.167 (0.3959) |  | 0.080 (0.4827) | 0.128 (0.3311)
  0.5 hours after dose |  |  |  |  | -0.514 (0.3729) |  | 0.131 (0.3518) | 0.384 (0.7434)
  1 hour after dose |  |  |  |  | -0.322 (0.6343) |  | 0.063 (0.2129) | -0.123 (0.3713)
  1.5 hours after dose |  |  |  |  | -0.353 (0.2722) |  | 0.109 (0.0729) | 0.375 (0.5060)
  2 hours after dose |  |  |  |  | -0.460 (0.2219) |  | 0.279 (0.5172) | 0.223 (0.3813)
  3 hours after dose |  |  |  |  | -0.263 (0.4014) |  | 0.016 (0.1550) | 0.435 (0.3796)
  5 hours after dose |  |  |  |  | -0.350 (0.7782) |  | 0.031 (0.2103) | -0.018 (0.6197)
  8 hours after dose |  |  |  |  | -0.454 (0.4568) |  | -0.028 (0.3062) | 0.271 (0.3849)

16. Other Pre Specified Outcome: EEG Parameter (DAY 12) - Gamma - Change From Baseline in Total Area of the Brain (Eyes Closed) - Consistent Change in Either Direction
Description: EEG parameter (DAY 12) - Gamma - Change from baseline in Total Area of the Brain (eyes closed) Cohort 5 & 7 , Cohort 6 did not reach Day 12; to identify a dose related change in EEG gamma bands to assess target engagement, a consistent change in either direction compared to placebo would be of interest
Time Frame: 8 hours after dose
Population: Safety population
Measure: Mean (Standard Deviation); unit: uV2
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 0 | 6 | 4
uV2
  Pre dose Day 12 |  |  |  |  | -0.075 (0.5040) |  | -0.065 (0.1789) | 0.015 (0.1749)
  0.5 hours post dose |  |  |  |  | -0.309 (0.7025) |  | -0.134 (0.2459) | 0.334 (0.3440)
  1 hours post dose |  |  |  |  | 0.193 (1.4967) |  | -0.107 (0.1970) | 0.253 (0.3448)
  1.5 hours post dose |  |  |  |  | 0.073 (0.9299) |  | -0.062 (0.1783) | 0.373 (0.3358)
  2 hours post dose |  |  |  |  | -0.207 (0.6381) |  | -0.087 (0.3025) | -0.046 (0.2830)
  3 hours post dose |  |  |  |  | -0.119 (0.6208) |  | -0.024 (0.2590) | 0.234 (0.3109)
  5 hours post dose |  |  |  |  | -0.506 (0.4329) |  | 0.040 (0.1775) | 0.090 (0.4258)
  8 hours post dose |  |  |  |  | 0.022 (1.0703) |  | -0.048 (0.0975) | 0.178 (0.2510)

ADVERSE EVENTS:
Time Frame: SAD cohorts 2 weeks, MAD cohorts up to 1 month
Description: From Day -1 (entry into unit) until 14 days after last dose (15 days for SAD cohorts and up to 29 days for MAD cohorts) note Mad Cohort 6, stopped due to randomisation error in pharmacy had 15 days of follow up for adverse events.
Arm/Group | AZD8108 20 mg SAD | AZD8108 60 mg SAD | AZD8108 95 mg SAD | Placebo SAD | AZD8108 50 mg MAD | AZD8108 90 mg MAD (6) | AZD8108 90 mg MAD (7) | Placebo MAD
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 6/6 | 4/6 | 4/6 | 3/6 | 3/6 | 1/8 | 4/6 | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8108 20 mg SAD (N=6) | AZD8108 60 mg SAD (N=6) | AZD8108 95 mg SAD (N=6) | Placebo SAD (N=6) | AZD8108 50 mg MAD (N=6) | AZD8108 90 mg MAD (6) (N=8) | AZD8108 90 mg MAD (7) (N=6) | Placebo MAD (N=4)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysguesia (Nervous system disorders) | 6 (6) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Halucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphoria (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Conversion of AZD8108 to active moiety AZD6567 was rapid, concentrations of AZD8108 were almost all below the level of quantification, no PK parameters were calculable for AZD8108 concentrations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days